CLINICAL TRIAL: NCT00584077
Title: Assessment of Cough Reflex in Lung Transplant Recipients
Status: Completed | Type: Observational
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Other Study IDs: 00-132
Record Dates: First submitted 2007-12-20; First posted 2008-01-02 (Estimated); Results first posted 2015-09-25 (Estimated); Last update posted 2018-11-02 (Actual); Status verified 2018-02

CONDITIONS: Complication of Transplanted Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Stable lung transplant recipients: All enrolled subjects receive the same procedures; bronchoscopy with administration of mechanical and chemical irritants to the airway mucosa

SUMMARY:
The purpose of this study is to evaluate the presence of cough reflex in the transplanted lung of patients who have had either a single or double lung transplant or heart-lung transplant at University of Texas Medical Branch. At the 1 year post transplant bronchoscopy, the presence of the cough reflex will be assessed by placing 3 to 5 ml of 5% dextrose and placement of the bronchial biopsy forceps on the airway mucosa. Three to four separate areas of the transplanted airways will be assessed. The cough reflex will be assessed by recording the surface electrical activity by placing external electrodes to monitor the movement of abdominal muscles during a cough. The data will be recorded and compared with recordings from coughs recorded using the surface electrical activity of a cough generated by non-transplant patients.

DETAILED DESCRIPTION:
Bronchoscopy Stable, lung transplant recipients undergoing surveillance bronchoscopy will be enrolled. We will exclude subjects with new or persistent cough, hypoxemia, new radiographic infiltrates, or hemodynamic instability.

Before bronchoscopy, patients will receive diazepam while codeine and atropine will be withheld. Upper airway anesthesia was performed using cotton swabs soaked with 4 % lidocaine applied on the oropharyngeal mucosa and gradually placed posteriorly with the aid of curved foreceps to anesthetize the supraglottic region. A trained individual will perform topical upper airway anesthesia over 15 minutes and adequate anesthesia will be determined once subjects fail to cough during foreceps application to the supraglottic region. Conscious sedation will be administered using intravenous midazolam while vital signs are monitored. Once adequate sedation is achieved, the bronchoscope will be introduced through the mouth beyond the vocal chords to the main carina and slowly advanced to the airway anastomosis. Coughing that occurs with advancement of the bronchoscope from the chords to the anastomosis will be addressed by maintaining the bronchoscope in an immobile neutral position for 60-180 seconds until coughing stops and the cough provocation will be performed.

Cough provocation Airway irritants will be applied in the following sequence: 1) one cm distal to anastomosis, 2) one cm proximal to anastomosis and 3) at the main carina. Chemical irritation will consist of 3 mL aliquots of 5 % dextrose water (D5W) instilled through the bronchoscope channel on the bronchial mucosa (21). Aliquots of D5W will be administered at each site on three separate occasions with a 60 second interval between administrations. Mechanical irritation will involve placement of the biopsy foreceps on the bronchial mucosa at each site. The sequence of airway irritation sites will always begin with the distal anastomosis followed by the proximal anastomosis and main carina.

Airway lidocaine administration Patients demonstrating a cough reflex at the distal anastomotic site will be recorded. After measurements are obtained at all airway sites, the bronchoscope will be reintroduced to the distal anastomosis and 3 mL of 4 % lidocaine instilled on the bronchial mucosa. Sixty seconds later, mechanical and chemical irritation of the proximal and distal anastomosis will be performed as previously outlined.

Cough assessment Cough frequency will be determined by counting audible coughs and abdominal muscle contractions measured with a surface electromyograph (EMG) recorder. Surface electrodes placed on the skin, 2 cm below each costal margin along the midclavicular line will be connected to an EMG recorder (Biopac Systems Inc, Santa Barbara, CA) linked to a dedicated computer. Continuous EMG recordings will be obtained 15 seconds before administration of the airway irritant to ensure absence of cough before airway irritant administration (Figure 1). Twenty seconds or more of recording will be obtained after airway irritant application. Cough will be defined as abdominal muscle contraction and audible expiratory sound.

ELIGIBILITY:
Inclusion Criteria:

* Lung transplant recipient
* Hemodynamically stable
* Capable of undergoing bronchoscopy

Exclusion Criteria:

* Pneumonia
* Hypoxemia (PaO2 < 70)
* Hemodynamic instability
* Coagulopathy
* Thrombocytopenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Single or double lung or heart-lung transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2000-04; Primary Completion 2006-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander G Duarte, MD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Duarte AG, Terminella L, Smith JT, Myers AC, Campbell G, Lick S. Restoration of cough reflex in lung transplant recipients. Chest. 2008 Aug;134(2):310-316. doi: 10.1378/chest.07-2934. Epub 2008 Mar 13. PMID 18339778

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects scheduled to undergo surveillance bronchoscopy were enrolled
Groups:
- Lung Transplant Recipients With Stable Lung Function: All enrolled subjects underwent bronchoscopy to determine presence of cough as well as the location of airway eliciting a cough response
Period: Overall Study
Arm/Group | Lung Transplant Recipients With Stable Lung Function
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lung Transplant Recipients With Stable Lung Function
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 49 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Coughs
Description: The number of coughs elicited by placement of biopsy forceps or instillation of dextrose solution on the airway mucosa. The presence of the cough reflex will be assessed with administration of mechanical (biopsy foreceps) and chemical (D5W) at the level of the main carina, proximal to airway anastomosis (native airway) and distal to the airway anastomosis (allograft airway).
Time Frame: 15-20 minutes
Measure: Mean (Standard Deviation); unit: Coughs
Arm/Group | Lung Transplant Recipients With Stable Lung Function
Number analyzed (Participants) | 15
Coughs | 7.3 (5.2)
Statistical Analysis 1: Comparison: Lung Transplant Recipients With Stable Lung Function; Each subject served as their own control as a comparison of the airway innervated (contralateral native lung) with the denervated airway (allograft); Test type: Superiority or Other; p < 0.01, ANOVA

2. Secondary Outcome: to Assess the Presence and Strength of the Cough Reflex in the Lower Airway for up to One Year
Description: Presence of cough as elicited by placement of biopsy forceps or instillation of dextrose solution on the airway mucosa. The presence of the cough reflex will be assessed with administration of mechanical (biopsy foreceps) and chemical (dextrose solution) at the level of the main carina, native lung airway and proximal and distal to the airway anastomosis. Lung transplant recipients underwent airway evaluations using the above protocel at 1.5 and 12 months after lung transplantation.
  after undergoing transplantation
Time Frame: 15-20 minutes
Population: Stable lung transplant recipients
Measure: Mean (Standard Deviation); unit: Coughs
Units Other Than Participants: Coughs
Groups:
- Lung Transplant Recipients With Stable Lung Function: All enrolled subjects underwent bronchoscopy to determine presence of cough as well as the location of airway eliciting a cough response. Subjects underwent bronchoscopy to elicit cough 1.5 months and 12 months after lung transplantation.
Arm/Group | Lung Transplant Recipients With Stable Lung Function
Number analyzed (Participants) | 8
Number analyzed (Coughs) | 24
Coughs
  Cough1.5 months with D5W at distal anastomosis | 0.63 (1.2)
  Cough 12 months with D5W at distal anastomosis | 7.3 (5.2)
  Cough1.5 months with foreceps atdistal anastomosis | 0.25 (0.46)
  Cough 12 months with foreceps atdistal anastomosis | 3.0 (2.3)
Statistical Analysis 1: Comparison: Lung Transplant Recipients With Stable Lung Function; For the cross-sectional and longitudinal groups, a comparison of cough frequency after airway irritation of the main carina, and the proximal and distal anastomotic sites was performed using one-way analysis of variance with Bonferroni test. In the longitudinal cohort, a comparison of the cough frequencies at different airway sites at 1.5 and 12 months was performed using one-way analysis of variance with Bonferroni test; Test type: Superiority or Other; p < 0.01, ANOVA — P value was adjusted for multiple comparisons using Bonferroni test

ADVERSE EVENTS:
Groups:
- Lung Transplant Recipients With Stable Lung Function: Enrolled subjects underwent bronchoscopy to assess for presence of cough reflex in the transpalnted and non-transplanted lung
Arm/Group | Lung Transplant Recipients With Stable Lung Function
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

LIMITATIONS AND CAVEATS:
The limitations of this trial are that the results apply to lung transplant recipients

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes